CLINICAL TRIAL: NCT02347436
Title: Effect of Transurethral Prostate Resection on 24 Hour Blood Pressure Measurement
Brief Title: Does Benign Prostatic Obstruction Cause Hypertension?
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/1117
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Prostatic Hyperplasia; Hypertension
Keywords: Transurethral Resection of Prostate
MeSH Terms: conditions — Prostatic Hyperplasia; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- benign prostatic hypertrophy: patients who are diagnosed with lower urinary tract symptoms caused by prostatic hypertrophy, undergo transurethral resection of the prostate, and post-surgery 24-hr ambulatory blood pressure measurement.
  Interventions: Procedure: 24-hr ambulatory blood pressure measurement
- inguinal hernia or hydrocele: patients who are diagnosed with lower urinary tract symptoms caused by inguinal hernia or hydrocele, undergo surgical inguinal hernia repair or hydrocele repair, and post-surgery 24-hr ambulatory blood pressure measurement
  Interventions: Procedure: 24-hr ambulatory blood pressure measurement

INTERVENTIONS:
Procedure: 24-hr ambulatory blood pressure measurement

SUMMARY:
The known correlation between benign prostatic hypertrophy (BPH) and hypertension could be explained by 3 theoretical pathway models. Whether hypertension causes BPH, BPH causes hypertension or the two are caused by a common factor is currently unknown.

In this study it will be investigated whether hypertension is due to the direct effects of infravesical obstruction to urinary outflow in patients with benign prostatic hyperplasia. The approach will be blood pressure measurement in patients who will have a resection of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Listed for inguinal hernia repair or hydrocele repair or transurethral resection of the prostate
* signed informed consent

Exclusion Criteria:

* Treatment with antihypertensive medication that has been started within 3 months of inclusion.
* Treatment with antihypertensive medication that has been started after inclusion and before final blood pressure measurements have been obtained 6 months after operation.
* Any reason that the investigator deems that the participant will not comply with follow-up.

Max Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on the waiting list for inguinal hernia repair, hydrocele operation, or transurethral resection of the prostate, at St Olavs University Hospital, Department of Surgery, Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
change in blood pressure | 7,5 months
  one measurement 6 weeks pre-surgery, and ambulatory measurement during 6 months post-surgery

SECONDARY OUTCOMES:
prostate symptom severity assessed by 'International prostate severity score' (questionnaire) | 7,5 months
  assessed by 'International prostate severity score' (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Carl-Jørgen Arum, md phd, Principal Investigator — St. Olavs University Hospital
Locations (1):
- St Olavs Hospital, Department of Urology, Trondheim, Norway